CLINICAL TRIAL: NCT02261805
Title: A Phase I/II Study of Ganetespib in Combination With Doxorubicin in Solid Tumors (Phase I) and Refractory Small Cell Lung Cancer (Safety Dose Expansion, Phase II)
Brief Title: A Phase I/II Study of Ganetespib in Combination With Doxorubicin
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company terminated drug support
Sponsor: Georgetown University (Other)
Collaborators: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-1195
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-03

CONDITIONS: Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasms; Small Cell Lung Carcinoma | interventions — STA 9090; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ganetespib and doxorubicin - Phase Ib Dose Level 1 (Experimental): Ganetespib 100 mg/m2 IV on days 1 and 8 of a 21-day cycle Doxorubicin 50 mg/m2 IV on day 1 of a 21-day cycle
  Interventions: Drug: Ganetespib; Drug: Doxorubicin
- Ganetespib and doxorubicin - Phase Ib Dose Level 2 (Experimental): Ganetespib 150 mg/m2 IV on days 1 and 8 of a 21-day cycle Doxorubicin 50 mg/m2 IV on day 1 of a 21-day cycle
  Interventions: Drug: Ganetespib; Drug: Doxorubicin
- Ganetespib and doxorubicin - Phase II Expansion (Experimental): Ganetespib 150 mg/m2 IV on days 1 and 8 of a 21-day cycle Doxorubicin 50 mg/m2 IV on day 1 of a 21-day cycle
  Interventions: Drug: Ganetespib; Drug: Doxorubicin

INTERVENTIONS:
Drug: Ganetespib
Drug: Doxorubicin
  Other Names: Adriamycin

SUMMARY:
This is a Phase I/safety dose expansion study of the combination of the drug ganetespib and doxorubicin in patients with advanced solid tumors. The purpose of the Phase I part of the study is to determine the recommended phase II dose of ganetespib when given in combination with doxorubicin. The recommended Phase II dose determined at the end of the dose escalation phase will be used to conduct a safety dose expansion phase in relapsed/refractory small cell lung cancer to determine if there is a signal of efficacy in this population.

DETAILED DESCRIPTION:
The dose escalation phase of the study will follow a standard 3+ 3 dose escalation scheme with two dose levels of ganetespib (1-- mg/m2 and 150 mg/m2) administered weekly on Days 1 and 8 of a 21-day cycle, in combination with a fixed dose of doxorubicin at 50 mg/m2 administered on Day 1 alone. After 4-6 cycles of combination therapy, continuation of single agent ganetespib will be permitted for subjects who are deriving clinical benefit.

Pharmacokinetic samples for plasma drug levels of ganetespib will be collected pre-dose and 4 hours after completion of treatment on Day 1 and Day 8 of cycle 1 only in subjects in the dose escalation phase.

The recommended Phase II dose determined at the end of the dose escalation phase will be used to conduct a safety dose expansion phase in relapsed/ refractory small cell lung cancer to determine if there is a signal of efficacy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation phase: histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. OR safety dose expansion phase: histologically or cytologically confirmed relapsed or refractory small cell lung cancer
* No more than 3 prior lines of chemotherapy; prior therapy with doxorubicin is permitted but no more than lifetime cumulative dose of 150 mg/m2; at least 3 weeks since prior chemotherapy or radiotherapy; at least 6 weeks if the last regimen included BCNU (1,3-bis(2-chloroethyl)-1-nitrosourea bis-chloronitrosourea) or mitomycin C
* Age >/= 18 years
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Life expectancy of greater than 3 months
* Adequate organ and marrow function
* Women of child-bearing potential must agree to avoid becoming pregnant and men must agree not to father a child for the duration of study participation.
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier.
* Receiving any other investigational agents
* Untreated symptomatic brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ganetespib or other agents used in the study
* Receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 or CYP2C18
* Left ventricular ejection fraction < 50%
* Known serious cardiac illness or medical conditions
* uncontrolled inter-current illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women
* HIV-positive on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Giaccone, MD PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Subramaniam DS, Liu SV, Crawford J, Kramer J, Thompson J, Wang H, Giaccone G. A Phase Ib/II Study of Ganetespib With Doxorubicin in Advanced Solid Tumors Including Relapsed-Refractory Small Cell Lung Cancer. Front Oncol. 2018 Mar 12;8:64. doi: 10.3389/fonc.2018.00064. eCollection 2018. PMID 29594044

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ganetespib and Doxorubicin - Phase Ib Dose Level 1 | Ganetespib and Doxorubicin - Phase Ib Dose Level 2 | Ganetespib and Doxorubicin - Phase II Expansion
Started | 3 | 6 | 2
Completed | 3 | 6 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ganetespib and Doxorubicin: Ganetespib 100 or 150 mg/m2 IV on days 1 and 8 of a 21-day cycle Doxorubicin 50 mg/m2 IV on day 1 of a 21-day cycle Ganetespib and doxorubicin
  Ganetespib and doxorubicin: IV ganetespib and doxorubicin
Arm/Group | Ganetespib and Doxorubicin
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The dose of ganetespib at which 1 or more out of 3-6 patients experiences a dose-limiting toxicity
Time Frame: 1 year
Measure: Number; unit: mg/m^2
Arm/Group | Ganetespib and Doxorubicin - Phase Ib Dose Level 1 | Ganetespib and Doxorubicin - Phase Ib Dose Level 2
Number analyzed (Participants) | 3 | 6
mg/m^2 | 100 | 150

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate included the count of confirmed complete responses (CR) and partial responses (PR) and was based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ganetespib and Doxorubicin - Phase Ib Dose Level 1 | Ganetespib and Doxorubicin - Phase Ib Dose Level 2 | Ganetespib and Doxorubicin - Phase II Expansion
Number analyzed (Participants) | 3 | 6 | 2
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Description: Adverse events were reported as pooling all subjects together and were not broken out by group.
Groups:
- Ganetespib and Doxorubicin: Ganetespib 100 or 150 mg/m2 IV on days 1 and 8 of a 21-day cycle Doxorubicin 50 mg/m2 IV on day 1 of a 21-day cycle
Arm/Group | Ganetespib and Doxorubicin
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganetespib and Doxorubicin (N=11)
Neutrophil count decreased (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ganetespib and Doxorubicin (N=11)
Constipation (Gastrointestinal disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 6 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Nausea (General disorders) | 8 (8)
Neutrophil count decreased (Immune system disorders) | 4 (4)
Pain (Nervous system disorders) | 2 (2)
Anorexia (General disorders) | 3 (4)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 2 (3)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Lymphocyte count decreased (Immune system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal anastomotic leak (Gastrointestinal disorders) | 1 (1)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Weight loss (Gastrointestinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 3 (3)
Hypophosphatemia (Blood and lymphatic system disorders) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1)
White blood cell decreased (Immune system disorders) | 1 (1)
AST elevation (Hepatobiliary disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Elavated LDH (Blood and lymphatic system disorders) | 1 (1)
Hypermagnesemia (Blood and lymphatic system disorders) | 1 (1)
Mucositis oral (Skin and subcutaneous tissue disorders) | 1 (1)
Back stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes